CLINICAL TRIAL: NCT01493921
Title: A Randomized, Double-Blind, Parallel, Vehicle-Controlled Phase III Trial to Assess the Efficacy and Safety of Topical SR-T100 Gel in the Treatment of Patients With Actinic Keratosis
Brief Title: Efficacy Study & Safety Evaluation of SR-T100 Gel in Actinic Keratosis Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: G&E Herbal Biotechnology Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GESRTAKA
Record Dates: First submitted 2011-12-15; First posted 2011-12-16 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Actinic Keratosis
Keywords: SR-T100 Clinical treatment against Actinic Keratosis; Actinic keratosis skin lesion treatment with SR-T100 gel; Skin lesion treatment with SR-T100 gel; SR-T100 gel treatment against skin lesion; Clinical efficacy study of SR-T100 gel
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SR-T100 gel (Experimental): Patient group receiving medication SR-T100 gel with active ingredient under investigation, enrolled subjects randomly assigned to this group to accurately depict statistical significance of the measured outcome.
  Interventions: Drug: SR-T100 gel
- Vehicle gel (Active Comparator): Patients given placebo with non-SR-T100 ingredients as they are being administered to patients, subjects are under random assignments from patient pool to depict statistically significant outcome measurement.
  Interventions: Drug: Vehicle gel

INTERVENTIONS:
Drug: SR-T100 gel — Patient will be instructed to self-apply approximately 0.3~0.5g of SR-T100 gel on 25 cm squared treatment area (avoiding the periocular areas, lips, and nares) once daily with an occlusive dressing for 16 weeks treatment period.
  Arms: SR-T100 gel
Drug: Vehicle gel — Patient wil be instructed to self-apply approximately 0.3~0.5g of vehicle gel (without active ingredient)per total of 25 cm squared treatment area (avoiding the periocular areas, lips, and nares) once daily with an occlusive dressing for 16 weeks treatment period.
  Arms: Vehicle gel

SUMMARY:
Studies of SR-T100 gel and its clinical relevance in the treatment of AK, providing adequate measured outcomes for skin lesion treatment. In addition to the high complete response rate (90.0%) as compared with the conventional therapy, the most significant result was that no undesirable side effects were associated with the use of SR-T100 gel. The result also shows approximately 80% of study subjects had a complete response in phase II clinical trial conducted in Taiwan; hence, result from our study model suggested SR-T100 gel offers beneficial therapeutic values in treatment of AK is harmless to the skin as well as high tolerance level displayed by majority of patients.

DETAILED DESCRIPTION:
The primary objective of this study is to demonstrate a clinically significant outcome involving SR-T100 topical gel developed against skin lesions such as AK. Furthermore, evaluation of SR-T100 efficacy & tolerability in treating AK lesions are developed as secondary objective in this clinical study. Patients with at least two clinically visible, discrete, non-hyperkeratotic, non-hypertrophic AK lesions on the arms, shoulder, chest, face and or scalp and at least one lesion of greater than or equal to 4mm in diameter within a total of 25 cm squared contiguous or non-contiguous treatment are expected to be enrolled. Candidate pool is then divided into two groups with random assignments of treatment group or placebo group. This randomization scheme will be generated by biostatistics and produced by a computer software program that incorporates a standard procedure for generating random probabilities. Study procedures include laboratory testings, analytical readings as well as clinical assessment practices for treatment efficacy and safety evaluations.

ELIGIBILITY:
Inclusion Criteria:

Male or female is 20 years of age or above and patient has at least two clinically visible, discrete, non hyperkeratotic, hypertrophic AK lesions located within a 25 cm squared contiguous or non contiguous treatment area including the arms, shoulder, chest, face and scalp. Patient has at least one histological confirmed actinic keratosis lesion of greater or equal to 4 mm in diameter within the selected treatment area.

Exclusion Criteria:

1. Patient has any dermatological disease and condition, such as atopic dermatitis, basal cell carcinoma, eczema, psoriasis, rosacea, squamous cell carcinoma, melanoma, or other possible confounding skin conditions in the treatment or surrounding area within 5cm distances from treatment area.
2. Patient had used the following treatments within 4 weeks prior to the study treatment initiation as immunomodulators or immunosuppressive therapy,interferon and cytotoxic drugs.
3. Patient treated with topical 5 FU, diclofenac gel, imiquimod, corticosteroids, retinoids, masoprocol on the treatment area within 4 weeks prior to the study treatment initiation.
4. Patient received cryodestruction, chemodestruction, curettage, photodynamic therapy, surgical excision on the treatment area within 4 weeks prior to the study treatment initiation.
5. Patient had received any of the following treatments on the treatment area in 6 months before study treatment initiation begins, such as psoralen plus UVA therapy, UVB therapy, laser abrasion, dermabrasion chemical peel.
6. Patient is known to be hypersensitive to the study medication.
7. Female who is pregnant, breast fed or considers of becoming pregnant while on the study.
8. Patient had used of any investigational drug within the past 30 days before enrollment.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2011-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Comparison of SR-T100 gel effect with those of vehicle gel (Placebo) on efficacy and tolerability in patients with actinic keratosis | 24 weeks
  The primary objective is to compare the complete clearance rate between treatment groups at 8 weeks after the completion of 16 weeks study treatment. The primary efficacy endpoint is to evaluate the complete clearance rate at 8 weeks after the completion of 16 weeks study treatment between treatment groups. The complete clearance is defined as the absence of visible or palpable AK lesions in the treatment area

SECONDARY OUTCOMES:
Evaluation of efficacy and tolerability of SR-T100 gel in AK treatment | 24 weeks
  SR-T100 clinical application in Actinic Keratosis treatment as direct proportional relationship to lesion size reduction, complete & partial clearance defined consequently as 100% & ≧75% reduction, coordinated toxicity & bio-safety reports supplements additional case study basis & foundation.

CONTACTS AND LOCATIONS:
Overall Officials: Hamm-Ming Sheu, MD, Principal Investigator — National Cheng-Kung University Hospital
Locations (6):
- Taiwan (6):
  - Chiayi Chang Gung Memorial Hospital, Chiayi City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Chi Mei Medical Center YongKang, Tainan
  - National Cheng Kung University Hospital, Tainan